CLINICAL TRIAL: NCT03151551
Title: A 52-Week Multicenter, Randomized, Open-Label, Parallel- Group Study Evaluating the Efficacy and Safety of Ixekizumab Versus Adalimumab in Patients With Psoriatic Arthritis Who Are Biologic Disease-Modifying Anti-Rheumatic Drug Naive
Brief Title: A Study of Ixekizumab (LY2439821) Versus Adalimumab in Participants With Psoriatic Arthritis
Acronym: SPIRIT-H2H
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16687; I1F-MC-RHCF (Other: Eli Lilly and Company); 2016-004585-25 (EudraCT Number)
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Results first posted 2019-04-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2019-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — ixekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental): 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline for all participants.
  80 mg ixekizumab given once every 2 weeks (Q2W) SC from week 2 to week 12 and once every 4 weeks (Q4W) thereafter for participants with moderate-to-severe plaque Ps.
  80 mg ixekizumab given SC Q4W starting week 4 for participants not meeting criteria for moderate-to-severe plaque Ps.
  Interventions: Drug: Ixekizumab
- Adalimumab (Active Comparator): 80 mg adalimumab given SC at baseline followed by 40 mg Q2W given SC starting week 1 for participants with moderate-to-severe plaque Ps.
  40 mg adalimumab given Q2W SC at baseline followed by 40 mg Q2W starting at Week 2 given SC for participants not meeting criteria for moderate-to-severe plaque Ps.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab
Drug: Adalimumab — Administered SC
  Arms: Adalimumab

SUMMARY:
The main purpose of this study is to evaluate the effectiveness and safety of ixekizumab versus adalimumab in participants with psoriatic arthritis (PsA) who are biologic disease-modifying anti-rheumatic drugs (DMARD) naive.

ELIGIBILITY:
Inclusion Criteria:

* Presence of established diagnosis of active psoriatic arthritis for at least 6 months, and currently meets Classification for Psoriatic Arthritis (CASPAR) criteria
* Active PsA defined as the presence of at least 3 (out of 68) tender and at least 3 (out of 66) swollen joints
* Presence of active plaque psoriasis with a BSA ≥3%
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* Have had an inadequate response when treated with 1 or more conventional synthetic disease-modifying antirheumatic drugs (csDMARDs)

Exclusion Criteria:

* Current or prior use of biologic agents for treatment of Ps or PsA
* Evidence of active inflammatory arthritic syndromes or spondyloarthropathies other than PsA
* Have participated in any study with interleukin 17 (IL-17) antagonists, including ixekizumab
* Serious disorder or illness other than psoriatic arthritis
* Serious infection within the last 3 months
* Active Crohn's disease or active ulcerative colitis
* Active vasculitis or uveitis
* Diagnosis of or history of malignant disease <5 years prior to randomization
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (131):
- Argentina (12):
  - Atencion Integral en Reumatología, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Clinica Adventista de Belgrano, Ciudad de Buenos Aires, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Instituto de Asist Reumatologica Integral, San Fernando, Buenos Aires
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Organizacion Medica de Investigacion - OMI, Ciudad Autonoma de Buenos Aire
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - Hospital Ramos Mejia, Ciudad Autonoma de Buenos Aire
  - Centro de Medicina Familiar Mindout Research, Ciudad Autonoma de Buenos Aire
  - CENUDIAB, Ciudad Autonoma de Buenos Aire
  - Consultora Integral de Salud S.R.L., Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER-San Juan, San Juan
- Australia (5):
  - Combined Rheumatology Practice (CRP), Kogarah, New South Wales
  - Rheumatology, The Queen Elizabeth Hospital, Woodville South, South Australia
  - Southern Clinical Research Pty Ltd, Hobart, Tasmania
  - Emeritus Research, Camberwell, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
- Austria (3):
  - Zentrum für klinische Studien Dr. Ursula Hanusch GmbH, Vienna
  - AKH, Vienna
  - Rheuma-Zentrum Wien Oberlaa, Vienna
- Belgium (5):
  - Reumaclinic, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Saint Joseph Hospital, Gilly
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Hopital Ambroise Pare, Mons
- Canada (5):
  - The Waterside Clinic, Barrie, Ontario
  - SKiN Center for Dermatology, Peterborough, Ontario
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Polmed Research Inc., Saskatoon, Saskatchewan
  - Group de recherche en maladies osseuses, Québec
- Denmark (2):
  - Frederiksberg Hospital, Frederiksberg, Capital Region
  - Aalborg Universitetshospital - Psykiatrien, Aalborg
- Finland (4):
  - Helsinki University Hospital, HYKS, Helsinki
  - Kiljava Medical Research, Hyvinkää
  - Terveystalo Kouvola, Kouvola
  - Turun Yliopistollinen Keskussairaala, Turku
- France (6):
  - Hôpital Trousseau, CHRU de Tours, Chambray-lès-Tours
  - Centre Hospitalier de Vendee Les Oudairies, La Roche-sur-Yon
  - Hopital Edouard Herriot, Lyon
  - Centre hospitalier universitaire Lapeyronie, Montpellier
  - Nouvel Hôpital Orléans La Source, Orléans
  - Hôpital Pierre-Paul Riquet, Toulouse
- Germany (4):
  - Klinikum der Universität München, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Rheumazentrum Ratingen, Ratingen, North Rhine-Westphalia
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (4):
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - UNO Medical Trials Kft., Budapest
  - Vital Medical Center, Veszprém
- India (13):
  - Care Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Panchshil Hospital, Ahmedabad, Gujarat
  - Byramjee Jeejeebhoy Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Shalby Hospital, Ahmedabad, Gujarat
  - Government Medical College & Sir Sayajirao General Hospital, Vadodara, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Narayana Hrudayalaya Hospital, Bangalore, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital &Medical Research Inst., Mumbai, Maharashtra
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Krishna Institute of Medical Sciences Ltd., Secunderabad, Telangana
  - Apollo Gleneagles Hospitals, Kolkata, West Bengal
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (7):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto Ortopedico Rizzoli, Bologna
  - Presidio Ospedaliero Vittorio Emanuele, Catania
  - Fondazione Universitaria degli Studi G D'Annunzio, Chieti
  - Policlinico di Tor Vergata, Roma
  - Complesso Integrato Columbus, Roma
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- Mexico (8):
  - CIMAB S.A. de C.V., Torreón, Coahuila
  - Centro Medico del Angel S.C., Mexicali, Estado de Baja California
  - Ctro Inv en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Grupo Médico CAMINO S.C., Mexico City, Mexico City
  - Clínica Enfermedades Crónicas y Procedimientos Especiales SC, Morelia, Michoacán
  - Centro Investigacion de Tratam Innovadores de Sinaloa SC, Culiacán, Sinaloa
  - Cemdeicy S.C.P., Mérida, Yucatán
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
- Antonius Ziekenhuis, Sneek, Netherlands
- Poland (5):
  - NZOZ Centrum Reumatologiczne Ind. Prak., Elblag
  - "Dermed" Centrum Medyczne Sp. z o.o., Lodz
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól
  - Rheuma Medicus Zakład Opieki Zdrowotnej, Warsaw
  - DermMEDICA Sp. z o.o., Wroclaw
- South Africa (9):
  - Greenacres Hospital, Port Elizabeth, Eastern Cape
  - Clinresco Centres (Pt) Ltd, Johannesburg, Gauteng
  - Suite 509 Umhlanga Netcare Medical Centre, Durban, KwaZulu-Natal
  - Arthritis Clinical Research Trial Unit, Pinelands, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
  - St Augustines Hospital, Durban
  - Emmed Research, Muckleneuk
  - Prof Ally, Pretoria
  - Suite 209A Jakaranda Hospital, Pretoria
- Spain (5):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, La Coruna
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Hospital Del Sagrado Coraz, Barcelona
  - Hospital Infanta Luisa, Seville
- Sweden (4):
  - Reumatologikliniken Västmanlands Sjukhus, Västerås, Västmanland County
  - Reumatologiska Kliniken Skånes universitetssjukhus Malmö, Malmo
  - Centrum för reumatologi, Stockholm
  - Reumatologiska Kliniken Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - HUG-Hôpitaux Universitaires de Genève, Geneva
- Ukraine (7):
  - Regional Clinical Hospital Center for Emergency medical care, Kharkiv
  - National Scientific Center "Strazhesko institute of cardio", Kyiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Multifield Medical Center of Odesa NMU (University Clinic#1), Odesa
  - Municipal Institution of Ternopil Regional Council, Ternopil
  - Vinnytsya Regional Clinical Hospital, Vinnytsia
  - Regional Clinical Hospital of Zaporizhzhia, Zaporizhzhia
- United Kingdom (12):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Royal Cornwall Hospital, Truro, Cornwall
  - Southampton General Hospital, Southampton, Hants
  - Wythenshawe Hospital, Wythenshawe, Manchester
  - Wishaw General Hospital, Wishaw, North Lanarkshire
  - Western General Hospital, Edinburgh, Scotland
  - Whipps Cross University Hospital, London, Surrey
  - North Tyneside General Hospital, North Shields, Tyneside
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - New Cross Hospital, Wolverhampton, West Midlands
  - St Lukes Hospital, Bradford, West Yorkshire
  - The Great Western Hospital, Swindon, Wiltshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Kristensen LE, McGonagle D, Rudwaleit M, Kameda H, Wurtzen PA, Ngantcha M, Holzkamper T, Smolen J. Synergistic Improvements in Synovitis, Enthesitis, and Patient-Reported Outcomes for Patients with Psoriatic Arthritis Treated with Ixekizumab in SPIRIT Trials. Rheumatol Ther. 2025 Apr;12(2):381-395. doi: 10.1007/s40744-025-00748-8. Epub 2025 Feb 27. PMID 40014255
- [Derived] Kirkham BW, Egeberg A, Behrens F, Pinter A, Merola JF, Holzkamper T, Gallo G, Ng KJ, Bolce R, Schuster C, Nash P, Puig L. A Comprehensive Review of Ixekizumab Efficacy in Nail Psoriasis from Clinical Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Rheumatol Ther. 2023 Oct;10(5):1127-1146. doi: 10.1007/s40744-023-00553-1. Epub 2023 Jul 3. PMID 37400681
- [Derived] Deodhar AA, Combe B, Accioly AP, Bolce R, Zhu D, Gellett AM, Sprabery AT, Burmester GR. Safety of ixekizumab in patients with psoriatic arthritis: data from four clinical trials with over 2000 patient-years of exposure. Ann Rheum Dis. 2022 Jul;81(7):944-950. doi: 10.1136/annrheumdis-2021-222027. Epub 2022 Apr 7. PMID 35393269
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Smolen JS, Sebba A, Ruderman EM, Schulze-Koops H, Sapin C, Gellett AM, Sprabery AT, Li L, de la Torre I, Gallo G, Liu-Leage S, Pillai S, Reis P, Nash P. Efficacy and Safety of Ixekizumab with or Without Methotrexate in Biologic-Naive Patients with Psoriatic Arthritis: 52-Week Results from SPIRIT-H2H Study. Rheumatol Ther. 2020 Dec;7(4):1021-1035. doi: 10.1007/s40744-020-00250-3. Epub 2020 Nov 16. PMID 33200394
- [Derived] Smolen JS, Mease P, Tahir H, Schulze-Koops H, de la Torre I, Li L, Hojnik M, Sapin C, Okada M, Caporali R, Gratacos J, Goupille P, Liu Leage S, Pillai S, Nash P. Multicentre, randomised, open-label, parallel-group study evaluating the efficacy and safety of ixekizumab versus adalimumab in patients with psoriatic arthritis naive to biological disease-modifying antirheumatic drug: final results by week 52. Ann Rheum Dis. 2020 Oct;79(10):1310-1319. doi: 10.1136/annrheumdis-2020-217372. Epub 2020 Jul 13. PMID 32660977
- See also: A Study of Ixekizumab (LY2439821) Versus Adalimumab in Participants With Psoriatic Arthritis (Spirit-H2H) — https://www.lillytrialguide.com/en-US/studies/psoriatic-arthritis/RHCF#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol and statistical analysis plan (SAP), the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Pre-assignment Details: Open-Label Treatment Period from Week 0 to Week 52 inclusive followed by Post-Treatment Follow-Up Period of up to a minimum of 12 weeks.
Groups:
- Ixekizumab: 160 milligrams (mg) ixekizumab (IXE) given subcutaneously (SC) at baseline for all participants.
  80 mg ixekizumab given once every 2 weeks (Q2W) SC from week 2 to week 12 and once every 4 weeks (Q4W) thereafter for participants with moderate-to-severe plaque Ps.
  80 mg ixekizumab given SC Q4W starting week 4 for participants not meeting criteria for moderate-to-severe plaque Ps.
  Follow-up: Participants did not receive drug during the Post-Treatment Follow-Up Period.
- Adalimumab: 80 mg adalimumab (ADA) given SC at baseline followed by 40 mg Q2W given SC starting week 1 for participants with moderate-to-severe plaque Ps.
  40 mg adalimumab given Q2W SC at baseline followed by 40 mg Q2W starting at Week 2 given SC for participants not meeting criteria for moderate-to-severe plaque Ps.
  Follow-up: Participants did not receive drug during the Post-Treatment Follow-Up Period.
Period: Open-Label Treatment Period
Arm/Group | Ixekizumab | Adalimumab
Started | 283 | 283
Received at Least One Dose of Study Drug | 283 | 283
IXE 160 mg at Baseline, 80 mg Q2W/Q4W | 49 | 0 (Row represents Ixekizumab data only.)
IXE 160 mg at Baseline, 80 mg Q4W | 218 | 0 (Row represents Ixekizumab data only.)
ADA 80 mg at Baseline, 40 mg Q2W | 0 (Row represents adalimumab data only.) | 51
ADA 40 mg at Baseline, 40 mg Q2W | 0 (Row represents adalimumab data only.) | 219
Completed | 265 | 259
Not Completed | 18 | 24
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 12 | 18
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Protocol Deviation | 1 | 2
Period: Post-Treatment Follow-Up Period
Arm/Group | Ixekizumab | Adalimumab
Started | 265 (All participants who received at least one dose of study drug could enter the follow-up period.) | 258 (All participants who received at least one dose of study drug could enter the follow-up period.)
Completed | 240 | 230
Not Completed | 25 | 28
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 20 | 22
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Groups:
- Ixekizumab: 160 milligrams (mg) ixekizumab (IXE) given subcutaneously (SC) at baseline for all participants.
  80 mg ixekizumab given once every 2 weeks (Q2W) SC from week 2 to week 12 and once every 4 weeks (Q4W) thereafter for participants with moderate-to-severe plaque Ps.
  80 mg ixekizumab given SC Q4W starting week 4 for participants not meeting criteria for moderate-to-severe plaque Ps.
- Adalimumab: 80 mg adalimumab (ADA) given SC at baseline followed by 40 mg Q2W given SC starting week 1 for participants with moderate-to-severe plaque Ps.
  40 mg adalimumab given Q2W SC at baseline followed by 40 mg Q2W starting at Week 2 given SC for participants not meeting criteria for moderate-to-severe plaque Ps.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab | Adalimumab | Total
Number analyzed (Participants) | 283 | 283 | 566
Age, Continuous [Median (Standard Deviation); unit: years] | 47.5 (12.02) | 48.3 (12.30) | 47.9 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 133 | 254
  Male | 162 | 150 | 312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 65 | 128
  Not Hispanic or Latino | 198 | 194 | 392
  Unknown or Not Reported | 22 | 24 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27 | 27 | 54
  Asian | 29 | 33 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 222 | 211 | 433
  More than one race | 5 | 11 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 31 | 27 | 58
  Hungary | 15 | 18 | 33
  Ukraine | 15 | 11 | 26
  United Kingdom | 13 | 7 | 20
  Switzerland | 1 | 3 | 4
  India | 20 | 26 | 46
  Spain | 24 | 18 | 42
  Canada | 5 | 5 | 10
  Sweden | 3 | 3 | 6
  Austria | 4 | 4 | 8
  Netherlands | 2 | 1 | 3
  Belgium | 6 | 5 | 11
  Finland | 5 | 6 | 11
  Poland | 24 | 29 | 53
  Denmark | 1 | 3 | 4
  Mexico | 32 | 33 | 65
  South Africa | 15 | 21 | 36
  Italy | 14 | 25 | 39
  Israel | 14 | 14 | 28
  Australia | 12 | 5 | 17
  France | 9 | 3 | 12
  Germany | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Simultaneously Achieving American College of Rheumatology 50 (ACR50) and Psoriasis Area and Severity Index 100 (PASI100)
Description: ACR50 response is a ≥50% improvement from baseline for tender joint count(TJC)& swollen joint count (SJC)& in at least 3 of the following 5 criteria: Participant's(pts) assessment of joint pain Visual Analog Scale (VAS),Pts Global Assessment of Disease Activity (PatGA)VAS, Physician's Global Assessment of Disease Activity (PGA)VAS, Pts assessment of physical function using the Health Assessment Questionnaire-Disability Index(HAQ-DI), or High Sensitivity(assay)C-Reactive Protein (hs-CRP). PASI is an index combining assessments of the extent of body-surface involvement in head, trunk, arms, legs, and severity of desquamation, erythema and plaque thickness in each region, yielding overall score of 0-no involvement, to 72-most severe involvement. Pts achieving PASI100 were defined as having 100% improvement in the PASI score compared to baseline. Pts with active plaque PsO with a BSA≥3% & PASI=0 at baseline were considered PASI100 responders if they had achieved PASI=0 & BSA=0 at week 24.
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants | 36 [30.4 to 41.6] | 27.9 [22.7 to 33.1]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; After data lock and initial analysis run, a medical inconsistency in baseline PASI data was identified (PASI=0 but BSA≥3%). The scenario was not anticipated or described in protocol or SAP. The inconsistency was resolved using medical judgment. The impacted participants had met baseline criteria for active psoriasis. Therefore, in the primary analysis, participants with baseline PASI=0 & BSA≥3% were considered PASI100 responders if, and only if, PASI=0 & BSA=0 achieved at week 24; Test type: Superiority; p = 0.036, Regression, Logistic; Rate Difference = 8.1, 95% CI 2-sided [0.5 to 15.8]

2. Secondary Outcome: Percentage of Participants Achieving ACR50
Description: ACR50 response is defined as a ≥50% improvement from baseline for tender joint count (TJC) and swollen joint count (SJC) and in at least 3 of the following 5 criteria: Participant's assessment of joint pain Visual Analog Scale (VAS), Participant's Global Assessment of Disease Activity (PatGA) VAS, Physician's Global Assessment of Disease Activity (PGA) VAS, participant's assessment of physical function using the Health Assessment Questionnaire-Disability Index (HAQ-DI), or High Sensitivity (assay) C-Reactive Protein (hs-CRP).
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants | 50.5 [44.7 to 56.4] | 46.6 [40.8 to 52.5]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Non-Inferiority — If the lower bound of the 2-sided 95% confidence Interval (CI) for the difference in proportions of responders on IXE minus ADA is greater than the pre-specified margin -12%, IXE will be deemed non-inferior to ADA; Rate Difference = 3.9, 95% CI 2-sided [-4.3 to 12.1]

3. Secondary Outcome: Percentage of Participants Achieving PASI100
Description: PASI is an index combining assessments of the extent of body-surface involvement in head, trunk, arms, legs, and severity of desquamation, erythema and plaque thickness in each region, yielding overall score of 0-no involvement, to 72-most severe involvement. Participants achieving PASI100 were defined as having 100% improvement in the PASI score compared to baseline. Any participants with active plaque psoriasis (PsO) with a BSA ≥3% and PASI = 0 at baseline were considered PASI100 responders if & only if they had achieved PASI=0 & BSA=0 at week 24.
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants | 60.1 [54.4 to 65.8] | 46.6 [40.8 to 52.5]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Regression, Logistic; Rate Difference = 13.4, 95% CI 2-sided [5.3 to 21.6]

4. Other Pre Specified Outcome: Change From Baseline in Tender Joint Count (TJC)
Description: TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model that included treatment group, concomitant conventional synthetic disease-modifying anti-rheumatic drugs (csDMARD) use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline TJC value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 239
score on a scale | -15.91 (0.566) | -14.88 (0.569)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.155, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-2.46 to 0.39], Standard Error of Mean 0.725

5. Other Pre Specified Outcome: Change From Baseline in Swollen Joint Count (SJC)
Description: SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS mean was calculated using MMRM model that included treatment group, concomitant conventional synthetic disease-modifying anti-rheumatic drugs (csDMARD) use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline SJC value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 239
score on a scale | -9.58 (0.196) | -9.53 (0.198)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.823, Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.54 to 0.43], Standard Error of Mean 0.249

6. Other Pre Specified Outcome: Change From Baseline in Participant's Assessment of Pain Visual Analogue Score (VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from Psoriatic arthritis (PsA) using a 100-millimeter(mm) horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by marking a vertical tick on the horizontal 100-mm scale, where the left end from 0 mm (no pain) to right end 100 mm (worst possible joint pain). LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline VAS value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 246
millimeters (mm) | -37.21 (1.623) | -36.54 (1.621)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.752, Mixed Models Analysis; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-4.80 to 3.47], Standard Error of Mean 2.104

7. Other Pre Specified Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity
Description: The patient's overall assessment of his or her PsA activity was recorded using a 100-mm horizontal VAS, where 0 represents no disease activity and 100 represents extremely active disease. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 246
Millimeter (mm) | -40.61 (1.594) | -37.82 (1.596)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.177, Mixed Models Analysis; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-6.83 to 1.26], Standard Error of Mean 2.060

8. Other Pre Specified Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The investigator was asked to give an overall assessment of the severity of the participant's current PsA activity using a 100-mm horizontal VAS, where 0 represents no disease activity and 100 represents extremely active disease. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 223 | 230
Millimeter (mm) | -48.15 (1.113) | -46.79 (1.097)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.332, Mixed Models Analysis; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-4.08 to 1.38], Standard Error of Mean 1.391

9. Other Pre Specified Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is the ACR Core Set laboratory measure of acute-phase reactant. It was measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on the participant's PsA. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline CRP value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: Milligram per Liter (mg/L)
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 234 | 238
Milligram per Liter (mg/L) | -5.68 (0.462) | -6.01 (0.461)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.592, Mixed Models Analysis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.86 to 1.50], Standard Error of Mean 0.599

10. Other Pre Specified Outcome: Change From Baseline in HAQ-DI
Description: HAQ-DI is a participant reported questionnaire that measures disease-associated disability (physical function). It consists of 24 questions with 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities. The disability section scores the participant's self-perception on the degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do), covering the 8 domains. The reported use of special aids or devices and/or the need for assistance of another person to perform these activities is assessed. The HAQ-DI is a composite ranging from 0-3 with lower scores indicating less functional disability. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline HAQ-DI value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 246
score on a scale | -0.68 (0.035) | -0.62 (0.035)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.15 to 0.03], Standard Error of Mean 0.045

11. Other Pre Specified Outcome: Percentage of Participants Simultaneously Achieving ACR50 and PASI100
Description: ACR50 response is a ≥50% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of VAS, Pts Global Assessment of Disease Activity (PatGA) VAS, Physician's Global Assessment of Disease Activity (PGA)VAS, participant assessment of physical function using the HAQ-DI, or High Sensitivity(assay) C-Reactive Protein (hs-CRP). PASI is an index combining assessments of the extent of body-surface involvement in head, trunk, arms, legs, and severity of desquamation, erythema and plaque thickness in each region, yielding overall score of 0-no involvement, to 72-most severe involvement. Participant achieving PASI100 were defined as having 100% improvement in the PASI score compared to baseline. Pts achieving PASI100 were defined as having 100% improvement in the PASI score compared to baseline. Pts with active plaque PsO with a BSA≥3% & PASI=0 at baseline were considered PASI100 responders if they had achieved PASI=0 & BSA=0 at week 52.
Time Frame: Week 52
Population: All randomized participants who had a baseline and at least one post-baseline ACR50 and PASI100 value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants | 39.2 [33.5 to 44.9] | 26.1 [21.0 to 31.3]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; After data lock and initial analysis run, a medical inconsistency in baseline PASI data was identified (PASI=0 but BSA≥3%). The scenario was not anticipated or described in protocol or SAP. The inconsistency was resolved using medical judgment. The impacted participants had met baseline criteria for active psoriasis. Therefore, in the primary analysis, participants with baseline PASI=0 & BSA≥3% were considered PASI100 responders if, and only if, PASI=0 & BSA=0 achieved at week 52; Test type: Superiority; p < 0.001, Regression, Logistic; Rate Difference = 13.1, 95% CI 2-sided [5.4 to 20.7]

12. Other Pre Specified Outcome: Change From Baseline in Disease Activity Score-CRP (DAS28-CRP)
Description: The DAS28-CRP is a measure of disease activity in 28 joints that consists of a composite numerical score with the following variables: TJC28, SJC28, hs-CRP (measured in milligrams per liter), and Participant's Global Assessment of Disease Activity recorded by participants on a 0 to 100 VAS. For DAS28-CRP, the Tender Joint Count 28 (TJC28) and Swollen Joint Count (SJC28) are a subset of TJC and SJC, and include 14 joints on each side of the body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. DAS28 values range from 0 to 9.4. Higher values indicate more severe symptoms and greater functional impairment. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline DAS28-CRP value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 226 | 228
score on a scale | -2.45 (0.071) | -2.36 (0.071)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.368, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.26 to 0.10], Standard Error of Mean 0.091

13. Other Pre Specified Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA)
Description: MDA is a composite of 7 key outcome measures: TJC ≤1; SJC ≤1; psoriasis activity and severity index (PASI total score) ≤1 or BSA ≤3; participant pain VAS score of ≤15; participant global disease activity VAS score of ≤20; HAQ-DI score ≤0.5; and tender entheseal points ≤1. Participants are classified as achieving MDA if they fulfill 5 of 7 outcome measures.
Time Frame: Week 52
Population: All randomized participants who had a baseline and at least one post-baseline MDA value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants
  MDA-6 Entheseal Points | 48.1 [42.2 to 53.9] | 42.8 [37.0 to 48.5]
  MDA-18 Entheseal Points | 47.3 [41.5 to 53.2] | 41.0 [35.3 to 46.7]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; MDA-18 Entheseal Points; Test type: Superiority; p = 0.108, Regression, Logistic; Rate Difference = 6.4, 95% CI 2-sided [-1.8 to 14.5]
Statistical Analysis 2: Comparison: Ixekizumab vs Adalimumab; MDA-6 Entheseal Points; Test type: Superiority; p = 0.179, Regression, Logistic; Rate Difference = 5.3, 95% CI 2-sided [-2.9 to 13.5]

14. Other Pre Specified Outcome: Percentage of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC)
Description: The PsARC is a composite criteria reported in terms of the percentage of participants achieving response according to the following criterion: TJC, SJC, PGA, and PatGA. Overall response is defined by improvement from baseline assessment in 2 of 4 criteria, 1 of which must be a joint count; there must not be worsening in any of the 4 criteria: at least 30% reduction in TJC, at least 30% reduction in SJC, at least a 20 millimeter (mm) reduction in PGA and at least a 20 mm reduction in PatGA.
Time Frame: Week 52
Population: All randomized participants who had a baseline and at least one post-baseline PsARC value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants | 66.8 [61.3 to 72.3] | 65.7 [60.2 to 71.3]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.846, Regression, Logistic; Rate Difference = -1.1, 95% CI 2-sided [-8.9 to 6.7]

15. Other Pre Specified Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI) Score
Description: The CPDAI is a validated instrument intended to assess composite psoriatic disease activity and response to therapy. Domains include peripheral arthritis as assessed by the number of tender and swollen joints and the HAQ-DI, skin as assessed by the PASI and the Dermatology Life Quality Index (DLQI), enthesitis as assessed by the number of sites with enthesitis and the HAQ-DI, and dactylitis as assessed by the number of digits affected. Each domain with the exception of spinal disease is scored from 0-3. Individual domain scores are summed to give an overall composite score (range 0-12) with a higher score indicating higher disease activity. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline CPDAI value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 237 | 234
score on a scale | -4.35 (0.136) | -3.85 (0.136)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.83 to -0.16], Standard Error of Mean 0.170

16. Other Pre Specified Outcome: Change From Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index in Participants With Enthesitis at Baseline
Description: The SPARCC enthesitis index evaluates tenderness in a total of 16 entheseal sites: the greater trochanter (right/left [R/L]), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial epicondyles of humerus (R/L),Lateral epicondyle humerus (R/L) and the supraspinatus insertion (R/L). Tenderness at each site is quantified on a dichotomous basis: 0 = nontender and 1 = tender. The results from each site are then added to produce a total score (range 0 to 16) with the Higher scores indicating more severe enthesitis. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline SPARCC score > 0. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 163 | 139
score on a scale | -3.93 (0.234) | -4.06 (0.241)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.687, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.48 to 0.72], Standard Error of Mean 0.305

17. Other Pre Specified Outcome: Change From Baseline in the Leeds Enthesitis Index (LEI) in Participants With Enthesitis at Baseline
Description: The LEI was developed specifically for use in PsA. It measures enthesitis at 6 sites (lateral epicondyle of humerus, right/left (R/L); medial femoral condyle,(R/L); Achilles tendon insertion, (R/L)). Each site is assigned a score of 0 (absent) or 1 (present); the results from each site are then added to produce a total score (range 0 to 6) with the higher scores indicating more severe enthesitis. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline enthesitis (LEI >0). Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 141 | 121
score on a scale | -1.93 (0.113) | -2.02 (0.116)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.507, Mixed Models Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.19 to 0.38], Standard Error of Mean 0.144

18. Other Pre Specified Outcome: Change From Baseline in the Leeds Dactylitis Index-Basic (LDI-B) in Participants With Dactylitis at Baseline
Description: The LDI-B measures the severity of dactylitis.In each digit,the ratio of the circumference(cf) of the affected digit to the cf of the digit on the opposite hand or foot measured in mm. Each dactylitic digit is defined by a minimum increase of 10% in cf over the contra-lateral digit.If the same digits on each hand or foot were thought to be involved,the clinician referred to a table of normative values for a value which was used to provide the comparison.If the ratio is >1.1,then subtract 1 from the calculated ratio and multiply it by 100 and the tenderness score of 0(not tender) or 1(tender).Otherwise,if the ratio of the cf of the digit is ≤1.1,then the LDI-B score is set to 0.LDI-B score can be >=0 with higher numbers indicating worse dactylitis.LS mean was calculated using MMRM model: treatment group,concomitant csDMARD use at baseline,moderate-to-severe Ps involvement,visit as fixed factors,baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline dactylitis (LDI-B >0). Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 35 | 47
score on a scale | -52.28 (11.495) | -48.89 (9.855)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.820, Mixed Models Analysis; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-32.78 to 25.99], Standard Error of Mean 14.951

19. Other Pre Specified Outcome: Change From Baseline in Psoriasis Body Surface Area (BSA)
Description: The investigator evaluates the percentage involvement of psoriasis on each participant's BSA on a continuous scale from 0% = no involvement to 100% = full involvement, where 1% corresponded to the size of the participant's handprint including the palm, fingers, and thumb. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline BSA value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 246 | 246
units on a scale | -12.33 (0.623) | -10.79 (0.613)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.052, Mixed Models Analysis; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-3.09 to 0.02], Standard Error of Mean 0.790

20. Other Pre Specified Outcome: Change From Baseline in the Nail Psoriasis Severity Index (NAPSI) Fingernails Score in the Subgroup of Participants With Fingernail Involvement at Baseline
Description: The NAPSI scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps by area of involvement. The fingernail is divided into quadrants. Each fingernail is given a score for fingernail bed Ps 0 (none) to 4 (Ps in 4 quadrants of the fingernail) and fingernail matrix Ps 0 (none) to 4 (Ps in 4 quadrants of the matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix Ps in each quadrant. The sum of all fingernails equals the total NAPSI score range is from 0 (no effect) to 80 (more severe psoriasis). LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had baseline fingernail involvement (NAPSI >0). Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 169 | 154
score on a scale | -17.78 (0.731) | -15.08 (0.742)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-4.57 to -0.84], Standard Error of Mean 0.949

21. Other Pre Specified Outcome: Change From Baseline in the Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from psoriasis is indicated by circling the number that best described the worst level of itching in the past 24 hours. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline NRS value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 242 | 246
score on a scale | -3.83 (0.159) | -3.54 (0.159)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.158, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.68 to 0.11], Standard Error of Mean 0.202

22. Other Pre Specified Outcome: Change From Baseline in Fatigue Severity NRS (Fatigue NRS) Score
Description: The Fatigue Severity NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine." Participants rate their fatigue (weariness, tiredness) by circling the 1 number that described their worst level of fatigue during the past 24 hours. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline Fatigue NRS value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 241 | 246
score on a scale | -3.03 (0.161) | -2.95 (0.161)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.711, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.49 to 0.33], Standard Error of Mean 0.21

23. Other Pre Specified Outcome: Change From Baseline in Medical Outcomes Study 36-item Short Form Health Survey (SF-36): Physical Component Summary (PCS)
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline PCS value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 240 | 246
score on a scale | 10.07 (0.526) | 9.55 (0.524)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.439, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.80 to 1.85], Standard Error of Mean 0.674

24. Other Pre Specified Outcome: Change From Baseline in SF-36: Mental Component Summary (MCS)
Description: as for outcome 23
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline MCS value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 240 | 246
score on a scale | 5.23 (0.660) | 4.77 (0.656)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.594, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-1.23 to 2.15], Standard Error of Mean 0.860

25. Other Pre Specified Outcome: Change From Baseline in Measures of Health Utility (EuroQol-5 Dimensions 5 Level [EQ-5D 5L]) United Kingdom(UK) Population-Based Index Score
Description: The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his/her current health state. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The descriptive part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The EQ-5D-5L health states were converted into a single summary index by applying a crosswalk using a UK Population value set to each of the levels in each dimension.This produced participant-level index scores between -0.594 and 1.0 (worse to better health). LS mean was calculated using MMRM model that included treatment group,concomitant csDMARD use at baseline,moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline EQ-5D 5L value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 240 | 245
score on a scale | 0.21 (0.013) | 0.21 (0.013)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.979, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.017

26. Other Pre Specified Outcome: Change From Baseline in Measures of Health Utility (EuroQol-5 Dimensions 5 Level [EQ-5D 5L]) VAS Score
Description: EQ-5D-5L is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his/her current health state using a 0 (worst health you can imagine) to 100mm VAS (best health you can imagine). LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: as for outcome 25
Measure: Least Squares Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 240 | 245
millimeters (mm) | 22.26 (1.37) | 17.48 (1.36)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 4.78, 95% CI 2-sided [1.28 to 8.28], Standard Error of Mean 1.782

27. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Scores range from 0 to 30 (less to more impairment), and a 4-point change from baseline is considered as the minimal clinically important difference threshold. LS mean was calculated using MMRM model that included treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit as fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interactions terms.
Time Frame: Baseline, Week 52
Population: All randomized participants who had a baseline and at least one post-baseline DLQI value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 241 | 246
score on a scale | -8.03 (0.273) | -6.91 (0.272)
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.78 to -0.46], Standard Error of Mean 0.335

28. Other Pre Specified Outcome: Percentage of Participants Answering "Mostly Satisfied" to Each Question in Treatment Satisfaction Questionnaire (TSQ)
Description: The TSQ is a clinician-administered questionnaire that provides an assessment of the patient's opinion of the effectiveness, safety, and overall satisfaction of the study medication. Participants were asked to respond to questionnaire items using a 4-point Likert scale (from "mostly satisfied" to "mostly dissatisfied").
Time Frame: Week 52
Population: All randomized participants who had a baseline and at least one post-baseline TSQ value. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
percentage of participants
  Effectiveness of Medication | 64.3 [58.7 to 69.9] | 58.7 [52.9 to 64.4]
  Effectiveness over Time of Medication | 62.9 [57.3 to 68.5] | 56.2 [50.4 to 62.0]
  Long Term Safety of Medication | 63.3 [57.6 to 68.9] | 58.7 [52.9 to 64.4]
  Overall Satisfaction with Medication | 64.0 [58.4 to 69.6] | 59.0 [53.3 to 64.7]
  Mostly Satisfied to any Questions | 70.0 [64.6 to 75.3] | 67.8 [62.4 to 73.3]
Statistical Analysis 1: Comparison: Ixekizumab vs Adalimumab; Effectiveness of Medication; Test type: Superiority; p = 0.165, Regression, Logistic; Rate Difference = 5.7, 95% CI 2-sided [-2.4 to 13.7]
Statistical Analysis 2: Comparison: Ixekizumab vs Adalimumab; Effectiveness over Time of Medication; Test type: Superiority; p = 0.098, Regression, Logistic; Rate Difference = 6.7, 95% CI 2-sided [-1.4 to 14.8]
Statistical Analysis 3: Comparison: Ixekizumab vs Adalimumab; Long Term Safety of Medication; Test type: Superiority; p = 0.241, Regression, Logistic; Rate Difference = 4.6, 95% CI 2-sided [-3.4 to 12.6]
Statistical Analysis 4: Comparison: Ixekizumab vs Adalimumab; Overall Satisfaction with Medication; Test type: Superiority; p = 0.215, Regression, Logistic; Rate Difference = 4.9, 95% CI 2-sided [-3.1 to 13.0]
Statistical Analysis 5: Comparison: Ixekizumab vs Adalimumab; Mostly Satisfied to any Questions; Test type: Superiority; p = 0.561, Regression, Logistic; Rate Difference = 2.1, 95% CI 2-sided [-5.5 to 9.7]

29. Other Pre Specified Outcome: Number of Participants Who Answered "Yes" to Any 10 Questions in Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a scale that captures the occurrence, severity, and frequency of suicide-related ideations and behaviors during the assessment period.
  1. Wish to be dead
  2. Non-specific active suicidal thoughts
  3. Active suicidal ideation with any methods (not plan) without intent to act
  4. Active suicidal ideation with some intent to act, without specific plan
  5. Active suicidal ideation with specific plan and intent
  6. Preparatory acts or behavior
  7. Aborted attempt
  8. Interrupted attempt
  9. Non-fatal suicide attempt
  10. Completed suicide
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab | Adalimumab
Number analyzed (Participants) | 283 | 283
Participants | 9 | 7

ADVERSE EVENTS:
Time Frame: Up To Week 52
Description: All participants who received at least one dose of study drug. Per protocol and statistical analysis plan, the primary and secondary analysis were performed to compare all ixekizumab participants together versus all adalimumab participants together. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly
Groups:
- Ixekizumab Follow-up; Adalimumab Follow-up: Follow-up: Participants did not receive drug during the Post-Treatment Follow-Up Period.
Arm/Group | Ixekizumab | Adalimumab | Ixekizumab Follow-up | Adalimumab Follow-up
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/283 | 0/265 | 0/260
Serious Adverse Events (participants affected / at risk) | 12/283 | 35/283 | 7/265 | 4/260
Other Adverse Events (participants affected / at risk) | 65/283 | 44/283 | 8/265 | 5/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab (N=283) | Adalimumab (N=283) | Ixekizumab Follow-up (N=265) | Adalimumab Follow-up (N=260)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/121 (0) | 1/133 (1) | 0/111 (0) | 0/123 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiologically isolated syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1/121 (1) | 0/133 (0) | 0/111 (0) | 0/123 (0)
Prostatitis (Reproductive system and breast disorders) | 0/162 (0) | 1/150 (1) | 0/154 (0) | 0/137 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (N=283) | Adalimumab (N=283) | Ixekizumab Follow-up (N=265) | Adalimumab Follow-up (N=260)
Injection site reaction (General disorders) | 16 (30) | 4 (9) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 38 (46) | 23 (26) | 5 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 18 (21) | 18 (23) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03151551/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT03151551/SAP_001.pdf